CLINICAL TRIAL: NCT05123885
Title: Impact Pronostique d'un événement Rythmique Ventriculaire Durant le Port de la LifeVest en Post-infarctus
Brief Title: Wearable Then Implantable Cardiac Defibrillator After Myocardial Infarction
Acronym: WICD-MI
Status: Completed | Type: Observational
Sponsor: Mathieu ECHIVARD (Other)
Responsible Party: Sponsor-Investigator, Mathieu ECHIVARD, Principal Investigator, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2021PI163
Record Dates: First submitted 2021-11-09; First posted 2021-11-17 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Infarction, Myocardial
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental:: Adult patients who benefited, between the start of 2015 and January 1, 2021, from a LifeVest after a myocardial infarction, followed by the implantation of an ICD before March 1, 2021.
  Interventions: Other: Study on Data

INTERVENTIONS:
Other: Study on Data — Study on Data

SUMMARY:
Sudden death from ventricular arrhythmia is a serious and common complication of myocardial infarction, especially with low left ventricular ejection fraction (LVEF). Implantable cardiac defibrillator (ICD) implantation is currently recommended at three months of optimal medical treatment in patients who have had a myocardial infarction and have a LVEF below 35%. This strategy indeed allows a reduction in mortality while early post-infarction implantation showed no benefit in terms of survival. However, the risk of sudden death at this period is the greatest and the temporary defibrillator vest, marketed under the name LifeVest, is now indicated in the early post-infarction period in patients with LVEF less than 35%. Indeed, the LifeVest would allow a reduction in sudden death of rhythmic origin in the first three months post-infarction. No study has yet investigated the prognostic significance of a ventricular rhythm disorder (ventricular tachycardia [VT] or ventricular fibrillation [VF]) occurring during this early and short (approximately 3 months) particular period of wearing the LifeVest: is this a random event, or is it an event predictive of a rhythmic recurrence? The aim of the study is to assess the association between the occurrence of a sustained ventricular rhythm disorder in the early post-infarction period, during the period of wearing the LifeVest (ventricular episodes detected, treated or not), and the risk of rhythmic recurrence at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who benefited, between the start of 2015 and January 1, 2021, from a LifeVest after a myocardial infarction, followed by the implantation of an ICD before March 1, 2021.

Exclusion Criteria:

* Patient opposition to the use of their data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who benefited, between the start of 2015 and January 1, 2021, from a LifeVest after a myocardial infarction, followed by the implantation of an ICD
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Rate of rhythmic recurrence defined as the occurrence of a sustained or treated ventricular rhythm disorder (VT or VF) during monitoring of the ICD. | 12 months after ICD implantation

SECONDARY OUTCOMES:
Rate of rhythmic recurrence defined as the occurrence of a sustained or treated ventricular rhythm disorder (VT or VF) during monitoring of the ICD. | Up to 7 years after ICD implantation
Rate of rhythmic storm defined by ACC / AHA / ESC 2006 guidelines (≥3 episodes of VF, sustained VT or appropriate shock in 24 hours). | 12 months and up to 7 years after ICD implantation]
Rate of need to set-up left ventricular assist device (LVAD) or heart transplantation. | : 12 months and up to 7 years after ICD implantation
Rate of all-cause death. | 12 months and up to 7 years after ICD implantation
Rate of hospitalization for heart failure worsening. | 12 months and up to 7 years after ICD implantation
Rate of rhythmic recurrence defined as the occurrence of a sustained or treated ventricular rhythm disorder (VT or VF) during monitoring of the ICD, and mortality from any cause. | Frame: 12 months and up to 7 years after ICD implantation
Rate of rhythmic recurrence defined as the occurrence of a sustained or treated ventricular rhythm disorder (VT or VF) during monitoring of the ICD, and mortality from any cause. | 12 months and up to 7 years after ICD implantation

CONTACTS AND LOCATIONS:
Locations (40):
- France (40):
  - Chu Amiens, Amiens
  - Ch D'Auxerre, Auxerre
  - Chu Besancon, Besançon
  - Polyclinique Reims-Bezannes, Bezannes
  - Chu Bordeaux Pessac, Bordeaux
  - Ch Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Chu Brest, Brest
  - Hospices Civils de Lyon, Bron
  - CHU de Caen, Caen
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Aphp Creteil, Créteil
  - Chu Dijon, Dijon
  - Clinique Essey Les Nancy, Essey-lès-Nancy
  - Chu Grenoble, La Tronche
  - Chu Lille, Lille
  - Chu Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Chu Aphm Marseille La Timone, Marseille
  - Hopital Prive Jacques Cartier, Massy
  - Chr de Metz Thionville, Metz
  - Chu Montpellier, Montpellier
  - Clinique Ambroise Pare, Nancy
  - Chu Nantes, Nantes
  - Chu Nimes, Nîmes
  - Chr D'Orleans, Orléans
  - Aphp Bichat, Paris
  - Php Hopital Europeen Georges Pompidou, Paris
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Ch de Roubaix, Roubaix
  - Chu Rouen, Rouen
  - Chu Aphp Salpetriere, Saint-Denis
  - Clinique Cardiologique Du Nord Saint-Denis, Saint-Denis
  - Chu Saint-Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Clinique Pasteur Toulouse, Toulouse
  - Chu Tours Saint-Avertin, Tours
  - Hopital Nord Franche-Comte, Trévenans
  - CHRU de Nancy, Vandœuvre-lès-Nancy